CLINICAL TRIAL: NCT03297021
Title: Effects of Ondansetron Dose and Timing on Rates of Post-operative Nausea and Vomiting
Brief Title: Effects of Ondansetron Dose and Timing on Post-operative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: GCO 17-1618
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Post-operative Nausea and Vomiting
Keywords: ambulatory surgery; post-operative nausea and vomiting; general anesthesia
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Random allocation by opaque envelope and random number generator. Investigator will draw up study medication and give to care-providers. Outcome assessor not present for drawing up of medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ondansetron 4mg Pre-emergence (Placebo Comparator)
  Interventions: Drug: Ondansetron 4 MG
- Ondansetron 8mg Pre-emergence (Experimental)
  Interventions: Drug: Ondansetron 8mg
- Ondansetron Pre-Incision and Pre-emergence (Experimental): 4mg Ondansetron Pre-Incision and 4mg Ondansetron Pre-emergence
  Interventions: Drug: Ondansetron 4 MG

INTERVENTIONS:
Drug: Ondansetron 4 MG — dose as per arm selection
  Arms: Ondansetron 4mg Pre-emergence; Ondansetron Pre-Incision and Pre-emergence
Drug: Ondansetron 8mg — dose as per arm selection
  Arms: Ondansetron 8mg Pre-emergence

SUMMARY:
The aim is to evaluate the effectiveness of three different regimens of prophylactic ondansetron on the incidence and severity of post-operative nausea and vomiting.

DETAILED DESCRIPTION:
Patients will be randomize to one of three arms: 4mg ondansetron pre-emergence, 8 mg ondansetron pre-emergence, or 4mg ondansetron pre-incision followed by 4mg ondansetron pre-emergence. Primary outcome will be incidence of PONV in the PACU prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II, III presenting for ambulatory surgery to be performed under general anesthesia

Exclusion Criteria:

* Patients with allergies or contraindications to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 165 patients assessed for eligibility 141 patients were randomized
Groups:
- Ondansetron 4mg Pre-emergence: Ondansetron 4 MG Pre-emergence
- Ondansetron 8mg Pre-emergence: Ondansetron 8mg Pre-emergence
Period: Overall Study
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
Started | 48 | 46 | 47
Completed | 43 | 42 | 43
Not Completed | 5 | 4 | 4
Not completed — Incomplete/illegible data sheet | 4 | 2 | 3
Not completed — Missing Post-Op Data | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence | Total
Number analyzed (Participants) | 43 | 42 | 43 | 128
Age, Continuous [Median (Full Range); unit: years] | 40 [33 to 51] | 39 [30 to 51] | 48 [31 to 57] | 40 [30 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 37 | 114
  Male | 2 | 6 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ASA Class [Median (Full Range); unit: units on a scale] — American Society of Anesthesiologist
  * ASA 1: A normal healthy patient.
  * ASA 2: A patient with a mild systemic disease.
  units on a scale | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
BMI [Median (Full Range); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 24.0 [21.0 to 27.0] | 25.0 [22.0 to 29.2] | 24.0 [21.0 to 28.6] | 24 [21 to 29.2]
History of PONV [Count of Participants; unit: Participants] — Post-operative nausea and vomiting
  Participants | 12 | 8 | 13 | 33
History of Vertigo [Count of Participants; unit: Participants] | 1 | 1 | 2 | 4
History of Motion Sickness [Count of Participants; unit: Participants] | 13 | 10 | 17 | 40
Current Smoker [Count of Participants; unit: Participants] | 3 | 0 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Nausea Scale
Description: Nausea Scale - full scale from 1-10, with higher score indicating more symptom of nausea
Time Frame: average of 4 hours in PACU and POD1
Population: only those participants with nausea completed the nausea scale
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
Number analyzed (Participants) | 10 | 7 | 8
score on a scale
  PACU | 3.5 [1.75 to 4.0] | 4.0 [3.0 to 6.0] | 4.0 [1.5 to 6.0]
  POD1: number analyzed (Participants) | 9 | 4 | 1
  POD1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 5.5] | 8.0 [8.0 to 8.0]

2. Secondary Outcome: Number of Participants With Episodes of Vomiting in the PACU
Description: Number of participants with episodes of vomiting in the Post Anesthesia Care Unit
Time Frame: average of 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
Number analyzed (Participants) | 43 | 42 | 43
Participants | 2 | 0 | 1

3. Secondary Outcome: Number of Participants With Symptoms on POD 1
Description: Number of participants with symptom presence of nausea or vomiting or headache on post-operative day one
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
Number analyzed (Participants) | 43 | 42 | 43
Participants
  Nausea | 9 | 4 | 1
  Vomiting | 1 | 1 | 0
  Headache | 5 | 5 | 3

4. Secondary Outcome: Number of Participants Who Needed Rescue Anti-emetics
Description: Number participants who needed rescue anti-emetics, i.e,, additional treatments needed to control nausea or vomiting in the PACU
Time Frame: average of 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
Number analyzed (Participants) | 43 | 42 | 43
Participants | 4 | 1 | 2

5. Secondary Outcome: Total Anesthesia Time
Time Frame: intraoperative, up to 3.5 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
Number analyzed (Participants) | 43 | 42 | 43
minutes | 116.0 [93.0 to 178.0] | 128.5 [86.5 to 186.25] | 118.0 [93.0 to 172.0]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Ondansetron 4mg Pre-emergence | Ondansetron 8mg Pre-emergence | Ondansetron Pre-Incision and Pre-emergence
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT03297021/Prot_SAP_000.pdf